CLINICAL TRIAL: NCT07288723
Title: Chronic Kidney Disease : Role of Biological Factors and Apolipoprotein L1 Encoding Gene
Brief Title: Chronic Kidney Disease : Role of Biological Factors and Apolipoprotein L1 Encoding Gene (APOL1)
Acronym: APOL1
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RNI_2018/03
Record Dates: First submitted 2025-11-14; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Diseases
Keywords: chronic kidney disease; stage renal disease; NT-ProBNP; FGF-23; APOL1 genetic variants
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A plasma bank, which will be used for the measurement of FGF-23 and DNA bank, which will be used for genotyping of APOL1 gene polymorphisms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case: Patients with stage 4 of chronic kidney disease (CKD)

SUMMARY:
Chronic kidney disease (CKD) is a major global public health issue. The present project focuses on the role of apolipoprotein L1 (APOL1) in patients with stage 4 CKD (glomerular filtration rate between 15 and 29 mL/min/1.73 m²).

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a worldwide public health problem. The project concerns the apolopoprotein L1 at stage 4 of severe chronic kidney disease (defined by a glomerular filtration rate of 29-15 ml / min / 1.73 m2).

Traditional risk factors (diabetes, cardiovascular diseases) and non-traditional such as inflammation and malnutrition are prognostic factors of mortality in our population.

Other parameters, less frequently described, would predict complications and mortality in patients on dialysis and in pre-dialysis the Fibroblast growth factor-23 (FGF-23) that regulates phosphates metabolism (Pereira, Juppner et al. 2009) and the " N terminal fragment of brain natriuretic peptide" (NT-proBNP), which plays a major role in regulation of blood pressure and extracellular volume.

Studies have suggested that black populations (African Americans) have a more rapid decline in kidney function than whites (European Americains).

The role of two variants (G1 and G2) of the gene encoding apolipoprotein L1 (APOL1) was mentioned. These APOL1 variants are common in African Americans (more than 50% are carriers of at least one risk allele). Carriers of 2 risk alleles would present a more rapid progression to end stage and, high-risk genotypes would explain most of the excess CKD risk for people of African descent. These variants of APOL1 Chronic kidney disease (CKD) is a worldwide public health problem. Our project concerns the apolopoprotein L1 at stage 4 of severe chronic kidney disease (defined by a glomerular filtration rate of 29-15 ml / min / 1.73 m2).

Traditional risk factors (diabetes, cardiovascular diseases) and non-traditional such as inflammation and malnutrition are prognostic factors of mortality in caribean population.

Other parameters, less frequently described, would predict complications and mortality in patients on dialysis and in pre-dialysis the Fibroblast growth factor-23 (FGF-23) that regulates phosphates metabolism and the " N terminal fragment of brain natriuretic peptide" (NT-proBNP), which plays a major role in regulation of blood pressure and extracellular volume.

Studies have suggested that black populations (African Americans) have a more rapid decline in kidney function than whites (European Americains). The role of two variants (G1 and G2) of the gene encoding apolipoprotein L1 (APOL1) was mentioned. These APOL1 variants are common in African Americans (more than 50% are carriers of at least one risk allele). Carriers of 2 risk alleles would present a more rapid progression to end stage and, high-risk genotypes would explain most of the excess CKD risk for people of African descent. These variants of APOL1 would also be associated with atherosclerotic cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 y and older, of both sexes, Afro Caribbeans
* Living in Guadeloupe
* Having been informed of objectives and constraints of the study and who have given their written consent.
* For patients with CKD : at stage 4 (GFR < than 30 ml / min / 1.73m2.), whatever the etiology of CKD, associated pathologies and treatments,
* For patients with normal renal function : serum creatinine < 10 mg/l.

Exclusion Criteria:

* Patients 18 y and older, of both sexes, Afro Caribbeans
* Living in Guadeloupe
* Having been informed of objectives and constraints of the study and who have given their written consent.
* For patients with CKD : at stage 4 (GFR < than 30 ml / min / 1.73m2.), whatever the etiology of CKD, associated pathologies and treatments,
* For patients with normal renal function : serum creatinine < 10 mg/l.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (≥18 years) with stage 4 chronic kidney disease (CKD), defined by a glomerular filtration rate (GFR) between 15 and 29 mL/min/1.73 m², patients are afro-caribeans and living i Guadeloupe. Participants will be recruited from a unique center (University Center Hospital of Guadeloupe) involved in the study.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2025-04-06 (Actual); Study Completion 2025-04-06 (Actual)

PRIMARY OUTCOMES:
Frequency of alleles (G1 and G2) of APOL1 | At baseline (study inclusion).
  The frequency of APOL1 risk alleles (G1 and G2 variants) will be determined in patients with stage 4 chronic kidney disease (CKD). This measure aims to describe the distribution of APOL1 genotypes within the study population and to identify the proportion of participants carrying one or two risk alleles, which may inform the analysis of associations with clinical and biochemical outcomes.
  Genotyping of APOL1 variants using DNA extracted from EDTA blood samples, analyzed by validated molecular biology techniques.

SECONDARY OUTCOMES:
Prevalence of Diabetes | At baseline (study inclusion)
  Percentage of participants with diabetes, defined according to ADA diagnostic criteria Measurement Method: Fasting glucose, HbA1c, and/or current antidiabetic treatment
Prevalence of Hypertension | At baseline (study inclusion)
  Percentage of participants with hypertension, defined according to ESC/ESH clinical criteria
  Unit of Measure: Percentage of participants
  Measurement Method: Standardized blood pressure measurement and/or current antihypertensive treatment
Prevalence of Malnutrition | At baseline (study inclusion)
  Percentage of participants meeting GLIM criteria for malnutrition
  Unit of Measure: Percentage of participants
  Measurement Method: BMI, serum albumin, weight loss history, clinical nutritional assessment
Echocardiographic Abnormalities | At baseline (study inclusion)
  Number of participants with at least one structural or functional cardiac abnormality (e.g., left ventricular hypertrophy, systolic or diastolic dysfunction)
  Unit of Measure: Number of participants
  Measurement Method: Standard transthoracic echocardiography (LVEF, E/e', wall thickness…)
Presence of Vascular Calcifications | At baseline (study inclusion)
  Percentage of participants with vascular calcifications detected on imaging.
  Unit of Measure: Percentage of participants
  Measurement Method: Imaging-based assessment (e.g., arterial calcium score according to clinical practice)
Plasma NT-proBNP concentration (pg/mL) | At baseline (study inclusion).
  Plasma concentration of N-terminal pro-B-type natriuretic peptide (NT-proBNP) measured by a validated immunoassay on blood samples collected at study inclusion. Higher NT-proBNP values reflect greater cardiac stress / volume overload. Results will be reported as continuous values (pg/mL) and summary statistics (mean, median, SD, IQR).
  Unit of Measure: pg/mL
Plasma Concentration of FGF-23 | At baseline (study inclusion)
  Plasma levels of Fibroblast Growth Factor-23 (FGF-23) will be measured in patients with stage 4 chronic kidney disease (CKD). The objective is to evaluate the association between circulating FGF-23 concentrations and APOL1 risk alleles (G1 and G2 variants), as well as to explore their potential relationships with cardiovascular and renal complications.
  FGF-23 concentrations will be quantified in plasma samples stored in the biobank using a validated immunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: Befa NOTO-KADOU-KAZA, MD, Principal Investigator — CHU de la Guadeloupe
Locations (1):
- CHU de la Guadeloupe, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No